CLINICAL TRIAL: NCT03499080
Title: Medication Free Treatment: Characteristics, Justification and Outcome
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Akershus (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Kristin Sverdvik Heiervang, Researcher Psychologist Phd, University Hospital, Akershus
Other Study IDs: medicationfree
Record Dates: First submitted 2018-03-23; First posted 2018-04-17 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Mental Illness
Keywords: Medication free treatment, mental illness, outcome
MeSH Terms: conditions — Mental Disorders | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients in medication free treatment: Inpatient unit dedicated to medication free treatment. This is an inpatient treatment unit for voluntary, planned treatment. The unit is staffed for a patient group that can be managed within a regime of open doors, voluntary treatment and low supervision. This means that high suicidal risk, severe acting out, active drug abuse etc. is excluded. They have an 8 week treatment program including Illness managment an recovery (IMR), Feedback informed treatment (FIT) and Affect consciousness treatment (ABT).
  Interventions: Behavioral: Medication free treatment
- Patients in treatment as Usual Åråsen: Inpatient unit colocated with the medication free unit. Same level of care. Similar treatment program, shorter treatment duration (on average 3 weeks).
  Interventions: Behavioral: Treatment as usual Åråsen
- Patients in treatment as Usual Myrvegen: Inpatient unit on a different location from the others. Same Level of care. Different treatment program. Intermediate treatment duration (mainly 4-6 weeks).
  Interventions: Behavioral: Treatment as usual Myrvegen

INTERVENTIONS:
Behavioral: Medication free treatment — Inpatient unit dedicated to medication free treatment. This is an inpatient treatment unit for voluntary, planned treatment. The unit is staffed for a patient group that can be managed within a regime of open doors, voluntary treatment and low supervision. This means that high suicidal risk, severe acting out, active drug abuse etc. is excluded. They have an 8 week treatment program including Illness managment an recovery (IMR), Feedback informed treatment (FIT) and Affect consciousness treatment (ABT).
  Groups: Patients in medication free treatment
Behavioral: Treatment as usual Myrvegen — Inpatient unit on a different location from the others. Same Level of care. Different treatment program. Intermediate treatment duration (mainly 4-6 weeks).
  Groups: Patients in treatment as Usual Myrvegen
Behavioral: Treatment as usual Åråsen — Unit colocated with the medication free unit. Similar treatment program. Short treatment duration (average 3 weeks).
  Groups: Patients in treatment as Usual Åråsen

SUMMARY:
In 2015 the Norwegian government, after initiative from user organizations, decided to implement medication free inpatient treatment units. The goal is to secure real options to medication for psychiatric illness, and to gather experiences with medication free options. Freedom of choice is a main concern.

The projects main aim is to study the outcome of medication free treatments of mental illness compared to treatment as usual, as well as characteristics of the treatment and the treatment population and why patients choose this treatment. Hereunder we aim to document who asks for these kinds of services and why, what kind of treatment they get, how they experience it, and how they respond to this kind of treatment. An important part will be to document whether the goal of increased freedom of choice between real treatment options is fulfilled.

Research questions

1. Does medication free treatment differ from treatment as usual? Are there any unique characteristics of the patient group who asks for this kind of treatment? What kind of treatment do they receive during their stay? How do they experience this treatment in comparison to treatment as usual? How is this in relation to the goals about increased freedom of choice? Does use of medication change during and/or after medication free treatment?
2. Why do patients choose medication free treatment? What are their reasons? What experiences lead to this wish?
3. What is the outcome of medication free treatment compared to treatment as usual?

DETAILED DESCRIPTION:
Background In 2015 the Norwegian government, after initiative from user organizations, decided to implement medication free inpatient treatment units. The goal is to secure real options to medication for psychiatric illness, and to gather experiences with medication free options. Freedom of choice is a main concern. (Aksjon for medisinfrie tilbud) The local unit under study DPS døgn Moenga at Akershus University Hospital has been given the assignment of developing a medication free treatment unit. This is an inpatient treatment unit for voluntary, planned treatment. High suicidal risk, severe acting out, active drug abuse etc. is excluded. The treatment program is 8 weeks long.

Status of knowledge The project has been controversial, especially with reference to the status of knowledge. Critiques have stated that the knowledge base for treating serious psychiatric disorders without medication is lacking (Gundersen, 2016; Røssberg, 2016). Concerns are raised about whether it can be harmful (Røssberg, 2016), whether it is necessary (Røssberg, Andreassen, & Malt, 2016) and whether it creates unfortunate dividing lines within health care (Røssberg et al., 2016). National guidelines recommend considering/offering medication for bipolar disorders, deep depression and psychosis (Helsedirektoratet, 2009, 2012, 2013). On the other hand, the knowledge base for use of psychotropic drugs is also being questioned, especially regarding long term effects (Bentall, 2009; Forand & DeRubeis, 2013; Moncrieff, 2009; Sohler et al., 2016; Whitaker, 2010/2014 (no), 2016). Studies on medication are amongst others criticized for not taking withdrawal effect sufficiently into account (Bentall, 2009; Forand & DeRubeis, 2013; Moncrieff, 2009; Whitaker, 2010/2014 (no), 2016). A randomized controlled study by Wunderink, Nieboer, Wiersma, Sytema, and Nienhuis (2013) indicates a follow up period of at least 3 years is necessary to see the benefits of drug reduction regarding antipsychotics.

Summing up, one can argue that generally, a considerable research base point to psychosocial treatment methods having an important place in the treatment of most psychiatric problems (Lambert, 2013; Wampold, 2001; Wampold & Imel, 2015). The more specific questions regarding pure psychosocial treatment for serious disorders and long term effects of psychotropic drugs are at least disputable, and probably under-researched.

Research questions

1. Does medication free treatment differ from treatment as usual? Patient characteristics, treatment received, experience, medication use.
2. Why do patients choose medication free treatment? What are their reasons? What experiences lead to this wish?
3. What is the outcome of medication free treatment compared to treatment as usual? Hypotheses The treatment outcome of medication free treatment is not inferior to treatment as usual.

Patients in medication free treatment will use less medication. Medication withdrawal may affect outcome in the short run.

Project methodology The design of the study is a mixed methods, observational design within a naturalistic treatment setting using qualitative and quantitative methods to address the research questions.

Moenga consist of two units, the medication free unit and a regular unit, which will be included for comparison. In addition we include a treatment unit on a different location for comparison; DPS Myrvegen. We aim for at least 200 n.

One complication is that this autumn it was decided that the units at Moenga shall move and reorganize sometime during 2018. This entail change of location, possible reorganizing of personnel and that the comparison unit at Moenga is joined with another inpatient unit at the new location. This may cause disruptions that can affect our results. We will study possible effects of this in our data, and may exclude parts of the gathered data and prolong the inclusion period.

We will collect survey data at start of treatment, weekly during treatment, at end of treatment (Work package 1), and at 6 months, 1 year, 2 years and 3 years follow up (work package 3). Register data will be collected 3 years back and 3 years follow up (work package 3). Patient interviews (work package 2) and personnel interviews (work package 4) are performed during spring 2018, the patient interviews near the end of the treatment stay. See measures for details.

Plan for data analyses Quantitative and qualitative analyses will be done according to the research questions. We will seek to compare the medication free unit and treatment as usual. Calculating propensity scores in the observational part of the study will be considered, to balance comparison groups (Austin, 2011).

Statistical power Exact power calculations are only possible in concrete, delimited statistical designs, and must necessarily be based on assumptions not always known before starting the study. In a design with 200 persons the total effect of one-way analysis of variance yield a statistical power of .80 for small to medium effect sizes. That is, the probability of detecting differences between groups will be .80 for effect sizes in the range .40 -.50. For pairwise comparisons between groups (with N=50), the probability of detecting effects in the range of Cohen's d >=. 40 will be about .80. In Cohen's pragmatic system, effect sizes with such magnitudes represent a "small to medium effect size". These estimations will also apply to change-scores between two points in time, given that the correlation between the two repeated measurements are r >= .5.

Study plan

Data collection:

Work package 1: Inclusion of patients for quantitative measurements starts April 2018 with a 12 months inclusion period. This may be prolonged if necessary.

Work package 2: Patient interviews will be performed during spring 2018. Work package 3: Follow up measures and register data will be collected until spring 2022.

Work package 4: Personnel interviews will be performed during spring 2018. Analysis Qualitative analyses will be performed within end of 2018. Quantitative analyses will start January 2019 Publishing Publishing of the results in scientific papers will take place mainly in 2019-2023.

Articles

1. "Medication free treatment: Does it differ from treatment as usual?" This article will address research question 1 and include qualitative data, Collaborate, BMQ, Inspire, CSQ-8, WAI, treatment received, use of medication and background data.
2. "Medication free treatment: Why?" This article will address research question 2 (Why do patients choose medication free treatment) and include qualitative data.
3. "Medication free treatment: Does it work?" This article will address the research questions and will include the outcome measures OQ-45, AII, Quality of life, HoNOs, GAF, CGI, drug use, diagnoses and register data. We will also look for correlations between use of medication and outcome, and therefore include measures of medication use.

Research group PhD Kristin S. Heiervang, head of the research group Quality and implementation in Mental Health Services at Akershus university hospital, is project manager (principal investigator) for the project.

Anders S. Wenneberg, specialist in clinical psychology, is the leader of the inpatient treatment facility. Wenneberg is also the project manager of the "Medication Free Treatment" at Akershus University Hospital, Moenga.

Ole André Solbakken is associate professor of clinical psychology and head of section at the Department of Psychology, University of Oslo.

Odd Arne Tjersland is professor of clinical psychology at the Department of Psychology, University of Oslo.

Jon T. Monsen is professor of clinical psychology at the Department of Psychology, University of Oslo.

Allan Abbass is professor, psychiatrist, and founding Director of the Centre for Emotions and Health at Dalhousie University in Halifax, Canada.

Kari Standal will be the PhD candidate. She is a psychologist at Akershus university hospital, specialized in adult treatment and psychotherapy (group treatment and affect consciousness).

Jill Arild, board member of "Mental Helse" and leader of the action group for medication free treatment is user represantive in the project.

Astrid Ringen Martinsen is a psychology student who will write her main thesis on the qualitative patient data.

Ingrid Engeseth Brakstad is a psychology student who will write her main thesis on the qualitative personnel data.

ELIGIBILITY:
Inclusion Criteria:

* Receiving planned treatment in the included treatment units
* Are able to fill out questionnaires in Norwegian with minimal help / be interviewed in norwegian
* Signed informed consent and willing to participate in the trial

Exclusion Criteria:

* Not able to fill out questionnaires or be interviewed in Norwegian.
* Beds dedicated acute crisis and usercontrolled beds

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with mental illness in the regions Øvre and Nedre Romerike who receive medication free treatment or treatment as usual at the same level of care (planned, voluntary inpatient treatment at DPS døgn) within the period from spring 2018 and 1-2 years forward, who are able to fill out forms / be interviewed in Norwegian and concent to participate.
Sampling Method: Non-Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Outcome Questionnaire-45 (OQ-45) | Filled out by patients at start of treatment, 1 time every week during the treatment program (typically 2 to 8 weeks), 1 time at end of treatment (typically at week 2-8) and at 6 months, 1 year, 2 years and 3 years
  This questionnaire was developed for tracking outpatients on a weekly basis. It measures symptom distress, interpersonal functioning and contentment with social role functioning, areas widely recognized as the essential ingredients of interest when assessing patient improvement. It is regarded suitable for patients with a wide range of diagnoses, sensitive to change over a short period of time, and brief and easy to administer (Lambert, Hansen, & Finch, 2001).

SECONDARY OUTCOMES:
The Working Alliance Inventory (WAI-SP) | Filled out by patients at start of treatment, 1 time every week during the treatment program (typically 2 to 8 weeks), 1 time at end of treatment (typically at week 2-8) and at 6 months, 1 year, 2 years and 3 years
  The WAI is one of the most widely used measures in research on working alliance and measures three aspects of the collaborative, purposive work in therapy: Bond, Task, and Goal. Research indicates that Bond, Task, and Goal represent the multidimensional construct working alliance is assumed to be (Horvath, 1994; ref. in Hersoug et al., 2009). WAI items are rated on a 7-point Likert-type scale ranging from 1 (never) to 7 (always), assessing the extent to which patient and therapist explicitly agree on the tasks and goals of therapy and the quality of the affective bond between them.
Beliefs about medicines questionnaire (BMQ) | Filled out by patients at start of treatment, end of treatment (typically at week 2-8) and at 6 months, 1 year, 2 years and 3 years
  The BMQ comprises two sections: the BMQ-Specific which assesses representations of medication prescribed for personal use and the BMQ-General which assesses beliefs about mcdicines in general. The pool of test items was derived from themes identified in published studies and from interviews with chronically ill patients. Principal Component Analysis (PCA) of the test items resulted in a logically coherent. 18 item, 4-factor structure which was stable across various illness groups. In this study we use the BMQ-Specific. The BMQ-Specific comprises two 5-item factors assessing beliefs about the necessity of prescribed medication (Specific-Necessity) and concerns about prescribed medication bascd on beliefs about the danger of dependence and long-term toxicity and the disruptive effects of medication (Specific-Concern).
INSPIRE measure of staff support for personal recovery | Filled out by patients at start of treatment, end of treatment (typically at week 2-8) and at 6 months, 1 year, 2 years and 3 years
  INSPIRE measure of staff support for personal recovery version 3 is included because the Recovery-tradition is a central part of the treatment program. Inspire has two subscales; Support and Relationship. The scale has demonstrated adequate psychometric properties (Williams et al., 2015).
CollaboRATE | Filled out by patients at start of treatment, end of treatment (typically at week 2-8) and at 6 months, 1 year, 2 years and 3 years
  Collaborate is a 3-item measure of shared decision making. CollaboRATE assesses three core SDM tasks: (1) explanation about health issues, (2) elicitation of patient preferences and (3) integration of patient preferences into decisions (Paul J. Barr et al., 2017). It has been found to have adequate psychometric properties in both simulated (Paul James Barr et al., 2014) and clinical (Paul J. Barr et al., 2017) settings.
The Client Satisfaction Questionnaire-8 (CSQ-8) | Filled out by patients at start of treatment, end of treatment (typically at week 2-8) and at 6 months, 1 year, 2 years and 3 years
  The Client Satisfaction Questionnaire-8 (CSQ-8) is an eight item questionnaire for measuring patient's global satisfaction with services. It has been shown to correlate well with the longer version, CSQ-18, and has shown good psychometric qualities regarding internal consistency, attendance, remainer-terminator status and greater client-reported symptomreduction (Attkisson & Zwick, 1982)
Affect Integration Inventory 42 (AII-42) | Filled out by patients at start of treatment, end of treatment (typically at week 2-8) and at 6 months, 1 year, 2 years and 3 years
  Affect Integration Inventory 42 (AII-42) is a short version of AII, a medium-length (112 items) self-rated assessment instrument that endeavors to measure capacities for experience and expression of nine affect states. These are important parts of the construct affect integration, the capacity to utilize affects for personal adjustment. A recent study has found satisfactory reliability, sound internal structure, and associations with external criteria, indicating good convergent and discriminant validity (Solbakken, Rauk, Solem, Lødrup, & Monsen, 2017).
Life satisfaction question | Filled out by patients at start of treatment, end of treatment (typically at week 2-8) and at 6 months, 1 year, 2 years and 3 years
  One question regarding life satisfaction from the project from the MANSA instrument (Clausen et al., 2015).
Questions regarding whether they specifically sought medication free treatment and why | Filled out by patients at start of treatment.
  Questions regarding whether they specifically sought medication free treatment and why (self-developed)
Background data | Filled out by patients at start of treatment.
  Sosiodemographic data, contact with family and network, caregiving, juridical information, health service use, health history, drug use, physical health, health history (from the project "Bedre psykosebehandling").
Treatment received | Filled out by patients at end of treatment (typically week 2-8).
  A form regarding what kind of treatment they have received during the stay, and benefit (adapted from Sintef Unimed, 2002)
Use of drugs | Filled out by patients at start of treatment, at 6 months, 1 year, 2 years and 3 years
  Use of drugs (questions from the project "Bedre psykosebehandling").
The Clinical Global Impressions Scale (CGI) | Filled out by clinician at start of treatment and end of treatment (typically week 2-8)
  The Clinical Global Impressions Scale (CGI) was developed for use in NIMH-sponsored clinical trials to provide a brief, stand-alone assessment of the clinician's view of the patient's global functioning prior to and after initiating a study medication (Guy, 1976; ref. in Busner & Targum, 2007) The CGI provides an overall clinician-determined summary measure that takes into account all available information, including a knowledge of the patient's history, psychosocial circumstances, symptoms, behavior, and the impact of the symptoms on the patient's ability to function. The CGI can track clinical progress across time and has been shown to correlate with longer, more tedious and time consuming rating instruments across a wide range of psychiatric diagnoses (Busner & Targum, 2007).
Health of the Nation Outcomes Scales (HoNOS) | Filled out by clinician at start of treatment and end of treatment (typically week 2-8).
  Health of the Nation Outcomes Scales (HoNOS) was developed to routinely measure outcomes for adults with mental illness. It is regarded adequate for assessing outcomes for different groups on a range of mental health-related constructs, and appropriate for routinely monitoring outcomes (Pirkis et al., 2005).
Global assessment of functioning (GAF) | Filled out by clinician at start of treatment and end of treatment (typically week 2-8).
  Global assessment of functioning (GAF) is one of the axes in the DSM diagnostic system from version III-R (Ullevål personlighetsprosjekt) until version 5. The multiaxial system was discarded in version 5 (Kress, Minton, Adamson, Paylo, & Pope, undated). From 1998 Statens helsetilsyn recommended all health institutions to use a minimum set of basic data ("minste basis datasett") which included a split version of GAF called S-GAF (Ullevål personlighetsprosjekt). The patient is ranged on two scales from 0-100 regarding symptoms and functioning. The psychometric properties of GAF are disputed (Kress et al., undated), but the measure is short, widely applied and mandatory in hospitals and therefore we include it.
Scale on alcohol (AUS) | Filled out by clinician at start of treatment and end of treatment (typically week 2-8).
  Scale on alcohol (AUS (Drake et al., 1990)
Scale on drugs (DUS) | Filled out by clinician at start of treatment and end of treatment (typically week 2-8).
  Scale on drugs (Mueser et al., 1995))
Diagnoses | Filled out by clinician at start of treatment and end of treatment (typically week 2-8).
  Diagnoses (including information on any diagnostic procedures used) (questions from the project "Bedre psykosebehandling").
Treatment received | Filled out by clinician at end of treatment (typically week 2-8).
  Treatment received (scheme adapted from SINTEF Helse, 2005).
Patient interviews | The interviews will be done close to the end of the treatment program (typically week 7).
  experience the treatment program, differences to other treatment they have been in and experience of freedom of choice regarding medication and other ways of coping. Interview guides will be developed by the phd candidate and a psychology student. The student will do pilot testing of the interview.
Register data | Register data will be documented at baseline, and at 6 months, 1 year, 2 years and 3 years follow up.
  We will seek approval and consent to get data from national official registers on health and use of health services (Norwegian Patient Register, HELFO for primary health and social care, NAV).
Staff interviews | The interviews are performed during spring 2018
  Interviews with staff on the medication free unit for exploring characteristics and differences to treatment as usual
Register data from the Medication Prescription Register | Collected at 3 years before treatment start, 2 years before, 1 year before, 6 months post treatment, 1 year post treatment, 2 years post treatment and 3 years post treatment
  Use of prescribed psychothropic medication
Questionnaire on medication filled out by patients | at start of treatment, at 6 monts, 1 year, 2 years and 3 years.
  Questionnaire regarding psychotrophic medication based on questions from the project "Bedre psykosebehandling"
Questionnaire on medication filled out by clinician | at start of treatment and end of treatment (typically at 2-8 weeks)
  Questionnaire regarding psychotrophic medication based on questions from the project "Bedre psykosebehandling"
Help with medication filled out by patient | at start of treatment, end of treatment (typically at 2-8 weeks) and at 6 months, 1 year, 2 years and 3 years.
  Help with medication: Questions developed in the project "Bedre psykosebehandling" about perceived quality of help and information regarding medication (Prosjekt Bedre psykosebehandling, n.d.).

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Heiervang, PhD, Principal Investigator — Akershus universitetssykehus
Locations (2):
- Norway (2):
  - DPS Øvre Romerike Døgn, Jessheim
  - DPS Nedre Romerike døgn, Lillestrøm

REFERENCES:
- [Background] Aksjon for medisinfrie tilbud. www.medisinfrietilbud.no. Retrieved from http://medisinfrietilbud.no
- [Background] Austin PC. An Introduction to Propensity Score Methods for Reducing the Effects of Confounding in Observational Studies. Multivariate Behav Res. 2011 May;46(3):399-424. doi: 10.1080/00273171.2011.568786. Epub 2011 Jun 8. PMID 21818162
- [Background] Benchimol EI, Smeeth L, Guttmann A, Harron K, Moher D, Petersen I, Sorensen HT, von Elm E, Langan SM; RECORD Working Committee. The REporting of studies Conducted using Observational Routinely-collected health Data (RECORD) statement. PLoS Med. 2015 Oct 6;12(10):e1001885. doi: 10.1371/journal.pmed.1001885. eCollection 2015 Oct. PMID 26440803
- [Background] Bentall, R. (2009). Doctoring the Mind. Why Psychiatric Treatments fail. London: Penguin Books.
- [Background] Forand, N. R., & DeRubeis, R. J. (2013). Combining medication and psychotherapyin the treatment of major mental disorders. In M. J. Lambert (Ed.), Bergin & Garfield's handbook of psychotherapy and behaviour change (6. ed., pp. 735-775). Hoboken, New Jersey: John Wiley & Sons inc.
- [Background] Gundersen, K. (2016). Medikamentfri psykiatri - eksperiment uten forskning. Aftenposten.
- [Background] Helse Sør-Øst. (2016). Overordnet protokoll for medisinfri behandling innen psykisk helsevern.
- [Background] Helsedirektoratet. (2009). Nasjonal retningslinje for diagnostisering og behandling av depresjon i primær- og spesialisthelsetjenesten. ( IS-1561).
- [Background] Helsedirektoratet. (2012). Nasjonal faglig retningslinje for utgreiing og behandling av bipolare lidingar (IS-1925). Helsedirektoratet.
- [Background] Helsedirektoratet. (2013). Nasjonal faglig retningslinje for utredning, behandling og oppfølging av personer med psykoselidelser ( IS-1957). Helsedirektoratet.
- [Background] Lambert, M. J. (2013). The efficacy and effectiveness of psychotherapy. In M. J. Lambert (Ed.), Bergin & Garfield's handbook of psychotherapy and behavior change (6. ed., pp. 169-219). Hoboken, New Jersey: John Wiley & sons, inc.
- [Background] Moncrieff, j. (2009). A straight talking Introduction to Psychiatric drugs. Herefordshire: PCCS Books.
- [Background] Røssberg, j. i. (2016, 13.06.16). Det er langt fra sikkert at det riktige er å innføre medisinfritt behandlingstilbud. Aftenposten.
- [Background] Røssberg, j. i., Andreassen, O. A., & Malt, U. (2016, 17.07.16). Medisinfrie tiltak for psykoselidelser er fortsatt et sjansespill. Aftenposten.
- [Background] Sohler N, Adams BG, Barnes DM, Cohen GH, Prins SJ, Schwartz S. Weighing the evidence for harm from long-term treatment with antipsychotic medications: A systematic review. Am J Orthopsychiatry. 2016;86(5):477-85. doi: 10.1037/ort0000106. Epub 2015 Dec 14. PMID 26652608
- [Background] Wampold, B. E. (2001). The Great Psychotherapy Debate. Models, Methods and Findings (2 ed.). Mahwah, New Jersey: Lawrence Erlbaum Associates publishers.
- [Background] Wampold, B. E., & Imel, Z. E. (2015). The Great Psychotherapy Debate. The Evidence for what makes Psychotherapy work (2 ed.). New York, London: Routledge, Taylor &Francis Group.
- [Background] Whitaker, R. (2010/2014 (no)). En psykiatrisk epidemi. Illusjoner om psykiatriske legemidler. Oslo: Abstract forlag.
- [Background] Whitaker, R. (2016). The case against antipsychotics. A review of their long-term effect. Weblog: Mad in America
- [Background] Wunderink L, Nieboer RM, Wiersma D, Sytema S, Nienhuis FJ. Recovery in remitted first-episode psychosis at 7 years of follow-up of an early dose reduction/discontinuation or maintenance treatment strategy: long-term follow-up of a 2-year randomized clinical trial. JAMA Psychiatry. 2013 Sep;70(9):913-20. doi: 10.1001/jamapsychiatry.2013.19. PMID 23824214
- [Derived] Standal K, Solbakken OA, Saltyte Benth J, Abbass A, Heiervang KS. Are People Worse Off in a Mental Health Treatment Paradigm Where Medication Is Deemphasised? A Naturalistic Noninferiority Trial of an Initiative to Improve Patient Choice. Int J Soc Psychiatry. 2025 Nov 23:207640251390930. doi: 10.1177/00207640251390930. Online ahead of print. PMID 41277153
- [Derived] Standal K, Solbakken OA, Rugkasa J, Halvorsen MS, Abbass A, Wirsching C, Brakstad IE, Heiervang KS. Medication-Free Treatment in Mental Health Care How Does It Differ from Traditional Treatment? Patient Prefer Adherence. 2024 Feb 3;18:315-335. doi: 10.2147/PPA.S435610. eCollection 2024. PMID 38327730